CLINICAL TRIAL: NCT02874703
Title: Mechanisms of Diastolic Dysfunction Among Persons With HIV Compared With Non-HIV Control Subjects
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: President and Fellows of Harvard College (Unknown); Nutrition Obesity Research Center at Harvard (Unknown)
Responsible Party: Principal Investigator, Tomas Neilan, MD, MD, Massachusetts General Hospital
Other Study IDs: 2015P000200
Record Dates: First submitted 2016-08-12; First posted 2016-08-22 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: HIV; Diastolic Dysfunction; Myocardial Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, plasma and serum

GROUPS / COHORTS (2):
- HIV-positive
  Interventions: Other: Cardiac MRI/MRS
- HIV-negative
  Interventions: Other: Cardiac MRI/MRS

INTERVENTIONS:
Other: Cardiac MRI/MRS

SUMMARY:
In this study, investigators plan to test two potential mechanisms contributing to diastolic dysfunction among asymptomatic persons with HIV who are on cART. The first proposed mechanism is that heightened systemic immune activation/inflammation in HIV contributes to myocardial inflammation, which in turn promotes myocardial fibrosis. The second mechanism is that ectopic fat deposition (increased visceral adiposity) in HIV relates to increased intramyocardial lipid content, which in turn contributes to diastolic dysfunction. Both HIV positive and HIV-negative participants will undergo cardiac MRI/ MRS imaging studies for evaluation of myocardial fibrosis, myocardial inflammation, and intramyocardial lipid content. Traditional markers of CVD risk, inflammatory markers/immune, hormonal markers, and markers of myocardial stretch/injury will be assessed in relation to cardiac MRI/MRS outcomes. Additionally, a small subset of participants with HIV will undergo longitudinal evaluations to assess effects of a clinically prescribed hormonal therapy on myocardial structure and function.

ELIGIBILITY:
HIV positive subjects

Inclusion Criteria:

* age ≥40 and ≤75 years
* documented HIV infection
* participant report that combination antiretroviral therapy (cART) (any regimen) has been taken stably without > 4 week interruption for at least 180 days prior to study entry (report of switching regimens in that time frame is permissible)

Exclusion Criteria:

* CD4 < 100 cell/mm3
* current active AIDS-defining illness
* current active or recent (not fully resolved within 30 days prior to study entry) systemic bacterial, fungal, parasitic, or viral infections (except HIV, HBV, human papillomavirus [HPV], or HCV)
* current active cancer
* clinical ASCVD, as defined by 2013 ACC/AHA guidelines (including previous diagnosis of AMI, ACS, stable or unstable angina, coronary or other arterial revascularization, stroke, TIA, PAD), by subject report
* clinical diagnosis of HFpEF or HFrEF, by subject report
* diagnosed DM on antihyperglycemic medication
* current, active use of immune suppressant medication including oral or intravenous corticosteroid or injectable biologic (oral ASA or NSAID use permitted)
* eGFR <45 ml/min/1.73 m2 calculated by CDK-EPI
* standard contraindications to MRI procedure based on MGH MRI Patient Procedure Screening Form - including history of severe allergy to gadolinium
* use of lipid lowering agents including statin drugs, fibrates, ezetimibe, red yeast rice, niacin or omega-3 fatty acids (>3 grams/day in standalone formulations) in the 90 days prior to study entry
* use of ACE inhibitor, ARB, or aldosterone receptor blocker in the 90 days prior to study entry
* pregnancy or breastfeeding (female subjects of reproductive potential)
* other medical, psychiatric, or psychological condition that, in the opinion of the study investigator, would interfere with completion of study procedures

HIV negative subjects:

Inclusion Criteria:

• age ≥40 and ≤75 years

Exclusion Criteria:

* HIV infection
* current active or recent (not fully resolved within 30 days prior to study entry) systemic bacterial, fungal, parasitic, or viral infections (except HIV, HBV, human papillomavirus [HPV], or HCV)
* current active cancer
* clinical ASCVD, as defined by 2013 ACC/AHA guidelines (including previous diagnosis of AMI, ACS, stable or unstable angina, coronary or other arterial revascularization, stroke, TIA, PAD), by subject report
* clinical diagnosis of HFpEF or HFrEF, by subject report
* diagnosed DM on antihyperglycemic medication
* current, active use of immune suppressant medication including oral or intravenous corticosteroid or injectable biologic (oral ASA or NSAID use permitted)
* eGFR <45 ml/min/1.73 m2 calculated by CDK-EPI
* standard contraindications to MRI procedure based on MGH MRI Patient Procedure Screening Form - including history of severe allergy to gadolinium
* use of lipid lowering agents including statin drugs, fibrates, ezetimibe, red yeast rice, niacin or omega-3 fatty acids (>3 grams/day in standalone formulations) in the 90 days prior to study entry
* use of ACE inhibitor, ARB, or aldosterone receptor blocker in the 90 days prior to study entry
* pregnancy or breastfeeding (female subjects of reproductive potential)
* other medical, psychiatric, or psychological condition that, in the opinion of the study investigator, would interfere with completion of study procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive and HIV negative participants
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Extracellular Volume (ECV), a measure of myocardial fibrosis on Cardiac MRI | 3 weeks

SECONDARY OUTCOMES:
Myocardial Inflammation on Cardiac MRI | 3 weeks
Intramyocardial fat on Cardiac MRI/MRS | 3 weeks
Diastolic function on Cardiac MRI | 3 weeks
Visceral Adiposity on MRI | 3 weeks
Inflammation/ immune markers | 3 weeks
Hormonal markers | 3 weeks
Markers of myocardial stretch | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Toribio M, Awadalla M, Drobni ZD, Quinaglia T, Wang M, Durbin CG, Alagpulinsa DA, Fourman LT, Suero-Abreu GA, Nelson MD, Stanley TL, Longenecker CT, Burdo TH, Neilan TG, Zanni MV. Cardiac strain is lower among women with HIV in relation to monocyte activation. PLoS One. 2022 Dec 30;17(12):e0279913. doi: 10.1371/journal.pone.0279913. eCollection 2022. PMID 36584183
- [Derived] Masenga SK, Romanelli A, Kooij KW. Plasma osteopontin in persons with HIV and the risk for cardiovascular disease. AIDS. 2023 Feb 1;37(2):355-357. doi: 10.1097/QAD.0000000000003445. No abstract available. PMID 36541647
- [Derived] Robinson JA, Toribio M, Quinaglia T, Awadalla M, Talathi R, Durbin CG, Alhallak I, Alagpulinsa DA, Fourman LT, Suero-Abreu GA, Nelson MD, Stanley TL, Longenecker CT, Szczepaniak LS, Jerosch-Herold M, Neilan TG, Zanni MV, Burdo TH. Plasma osteopontin relates to myocardial fibrosis and steatosis and to immune activation among women with HIV. AIDS. 2023 Feb 1;37(2):305-310. doi: 10.1097/QAD.0000000000003417. Epub 2022 Nov 3. PMID 36541642
- [Derived] Toribio M, Fulda ES, Chu SM, Drobni ZD, Awadalla M, Cetlin M, Stanley TL, North CM, Nelson MD, Jerosch-Herold M, Szczepaniak LS, Burdo TH, Looby SE, Neilan TG, Zanni MV. Hot Flashes and Cardiovascular Disease Risk Indices Among Women With HIV. Open Forum Infect Dis. 2021 Jan 12;8(2):ofab011. doi: 10.1093/ofid/ofab011. eCollection 2021 Feb. PMID 33575428
- [Derived] Toribio M, Awadalla M, Cetlin M, Fulda ES, Stanley TL, Drobni ZD, Szczepaniak LS, Nelson MD, Jerosch-Herold M, Burdo TH, Neilan TG, Zanni MV. Brief Report: Vascular Dysfunction and Monocyte Activation Among Women With HIV. J Acquir Immune Defic Syndr. 2020 Oct 1;85(2):233-238. doi: 10.1097/QAI.0000000000002419. PMID 32541385
- [Derived] Zanni MV, Awadalla M, Toribio M, Robinson J, Stone LA, Cagliero D, Rokicki A, Mulligan CP, Ho JE, Neilan AM, Siedner MJ, Triant VA, Stanley TL, Szczepaniak LS, Jerosch-Herold M, Nelson MD, Burdo TH, Neilan TG. Immune Correlates of Diffuse Myocardial Fibrosis and Diastolic Dysfunction Among Aging Women With Human Immunodeficiency Virus. J Infect Dis. 2020 Mar 28;221(8):1315-1320. doi: 10.1093/infdis/jiz184. PMID 31100122